CLINICAL TRIAL: NCT06673498
Title: Lusutrombopag Combined With Recombinant Human Thrombopoietin for the Treatment of Thrombocytopenia in Patients With Chronic Liver Disease Destined to Undergo Elective Invasive Surgery: a Prospective, Multicentre, Single-arm Clinical Study
Brief Title: Lusutrombopag Combined With Recombinant Human Thrombopoietin for the Treatment of Thrombocytopenia in Patients With Chronic Liver Disease Destined to Undergo Elective Invasive Surgery
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Anhui Provincial Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024KY402
Record Dates: First submitted 2024-10-27; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Thrombocytopenia
MeSH Terms: conditions — Thrombocytopenia | interventions — Thrombopoietin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): Lusutrombopag combined with recombinant human thrombopoietin
  Interventions: Drug: Lusutrombopag combined with recombinant human thrombopoietin

INTERVENTIONS:
Drug: Lusutrombopag combined with recombinant human thrombopoietin — After eligibility is confirmed, patients will begin treatment with Lusutrombopag +recombinant human thrombopoietin on Day 1, and study treatment will continue for 7 days

SUMMARY:
To assess the efficacy and safety of lusutrombopag combined with recombinant human thrombopoietin for the treatment of thrombocytopenia in patients with chronic liver disease destined to undergo elective invasive surgery.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand the study and willingness to comply with all study procedures by voluntarily signing an informed consent form prior to screening.
* Male or female, 18 years of age or older at the time of signing the informed consent form.
* Patients with chronic liver disease.
* Baseline platelet count ≤ 35 x 109/L prior to enrolment on day 1.
* Proposed elective invasive surgery that meets the following conditions: - Platelet transfusion may be required - Expected to be performed between days 9 and 15 after enrolment - Excludes extremely high-risk surgical operations such as open abdomen, open chest, open skull, and direct cardiac surgery.
* Eastern Collaborative Oncology Group (ECOG) Physical Status (PS) score of 0 or 1.
* According to the researcher, it will be able to fulfil the requirements of this study.
* Male patients who are infertile or who agree to use adequate contraception (including the use of condoms containing spermicides) from the start of screening until completion of the post-treatment phase.
* Female patients who are not menopausal or surgically sterilised need to agree to the use of highly effective contraception (including implants, injectable contraception, combined hormonal contraception [including vaginal rings], intrauterine devices, or partner-performed vasectomies) from the start of the screening until the completion of the end-of-treatment phase. The use of barrier contraception with or without spermicide, double barrier contraception and oral contraceptives alone is not adequate.

Exclusion Criteria:

* Presence of any of the following diseases: - Haematopoietic tumours - Aplastic anaemia - myelodysplastic syndrome - myelofibrosis - Congenital thrombocytopenia - Drug-induced thrombocytopenia - Immune thrombocytopenia - Systemic infections requiring treatment, except viral hepatitis
* Any solid malignancy with the following conditions: - Patients will require systemic chemotherapy, targeted therapy, immunotherapy, traditional herbal medicine or radiotherapy for that malignancy during the study period - Malignancy with lymph node metastasis, distant metastasis or peripheral organ invasion - Exceptions are: - Malignancy is a therapeutic target for the first invasive surgery - Non-melanoma skin cancers, intramucosal cancers, or carcinoma in situ that do not require any treatment during the study period.
* History of liver transplantation.
* Previous or current thrombosis or pre-thrombotic state (e.g., cerebral infarction, cardiac infarction, angina pectoris, coronary stenting, angioplasty, coronary artery bypass grafting, congestive heart failure [New York Heart Association {NYHA} class III/IV], cardiac arrhythmia [e.g., atrial fibrillation] known to increase the risk of thromboembolic events, pulmonary thromboembolism, deep venous thrombosis, or disseminated vascular (intravascular coagulation syndrome).
* Presence of any of the following conditions at screening: - Symptoms of hepatic encephalopathy with Child-Pugh Hepatic Encephalopathy Score 3 (occasional coma), with or without treatment for hepatic encephalopathy - Ascites uncontrolled by medications - Total bilirubin > 3 mg/dL
* Presence of history or evidence of a disease with bleeding risk (e.g. coagulation factor deficiency or vascular haemophilia factor vWF deficiency).
* History or evidence of any of the following disorders: - Congenital thrombophilia (e.g., antithrombin deficiency, protein C deficiency, protein S deficiency, or coagulation factor [coagulation factor V Leiden] mutation) - Acquired thrombophilia (e.g., antiphospholipid antibody syndrome, paroxysmal nocturnal haemoglobinuria, hyperhomocysteinemia, or elevated coagulation factor VIII) - Budd-Chiari syndrome
* Portal vein tumour embolism.
* Ultrasound, computed tomography (CT) or magnetic resonance imaging (MRI) within 28 days prior to enrolment showing portal vein thrombosis, or a history of portal vein thrombosis.
* Upper gastrointestinal endoscopy within 180 days prior to enrolment showing bleeding due to untreated gastro-oesophageal varices or the need to undergo treatment (except for patients in whom the first invasive procedure was performed to treat gastro-oesophageal varices).
* Prior to enrolment, the bleeding score was ≥ grade 2 according to the World Health Organization (WHO) Bleeding Scale.
* Use of any of the following medications or treatments within 90 days prior to enrolment: - Antineoplastic agents, excluding transcatheter arterial chemoembolisation (TACE) and oil iodide embolisation - Interferon agents - Radiotherapy - Radiotherapy - Any experimental drug
* Known hypersensitivity to the test drug or any of its excipients.
* Positive human immunodeficiency virus antigen/antibody test at screening.
* Women who are pregnant or breastfeeding.
* Patients deemed ineligible by the investigator for any other reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-11-10 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of respondents at day 8 | Day 8
  Responders were defined as subjects who achieved a platelet count of ≥50 × 10^9/L and an increase of ≥20 × 10^9/L from baseline and who did not receive emergency treatment for bleeding

SECONDARY OUTCOMES:
Proportion of subjects achieving a platelet count ≥50 × 10^9/L on or after day 8 and within 2 days prior to elective invasive surgery | on or after day 8 and within 2 days prior to elective invasive surgery
  Proportion of subjects achieving a platelet count ≥50 × 10^9/L on or after day 8 and within 2 days prior to elective invasive surgery
Proportion of subjects meeting the definition of responder at any time during the study period | Each routine blood test on or after day 8
  Responders were defined as subjects who achieved a platelet count of ≥50 × 10^9/L and an increase of ≥20 × 10^9/L from baseline and who did not receive emergency treatment for bleeding
Proportion of subjects requiring emergency treatment for bleeding at any time during the study period | During the procedure
  Proportion of subjects requiring emergency treatment for bleeding at any time during the study period
Number and dose of platelet transfusions during the study period | During the procedure
  Number and dose of platelet transfusions during the study period

CONTACTS AND LOCATIONS:
Overall Officials: Lianxin Liu, Principal Investigator — Anhui Provincial Hospital
Locations (2):
- China (2):
  - No.2 People's Hospital of Fuyang city, Fuyang, Anhui
  - Anhui province hospital, Hefei, Anhui

IPD SHARING:
Plan to Share IPD: No